CLINICAL TRIAL: NCT06788795
Title: Clinical Effectiveness of a Wearable Hydration Device
Brief Title: Effectiveness of a Wearable Hydration Device
Acronym: DRINK
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Joseph Piktel, Associate Professor, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00000196; R42AG080886 (NIH)
Record Dates: First submitted 2024-12-11; First posted 2025-01-23 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Dehydration; Syncope and Collapse
Keywords: dehydration; total body water; bioimpedence; emergency department
MeSH Terms: conditions — Dehydration; Syncope; Emergencies

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: Device and phones are identical but apps will either prompt or not prompt
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Device with Interactive Phone App (Active Comparator): In this arm, patients will receive the wearable dehydration device and receive the phone app, which will include prompts to check their dehydration status and to drink more fluids if necessary
  Interventions: Device: Device with Phone App
- Device without Interactive Phone APp (Sham Comparator): In this arm, patients will receive the wearable dehydration device without the phone app
  Interventions: Device: Device without Phone App

INTERVENTIONS:
Device: Device with Phone App — This is the intervention where the patients will be given both the wearable dehydration device as well as the phone app
  Arms: Device with Interactive Phone App
Device: Device without Phone App — This is the intervention where the patients will receive the device alone
  Arms: Device without Interactive Phone APp

SUMMARY:
Dehydration among older adults a costs billions of dollars in US healthcare every year because no robust solution exists to detect changes in hydration and prevent negative outcomes. In this project, TritonX Technologies Inc. and academic research partners plan to test whether a newly created wearable sensor that measures hydration in real time can promote hydration and prevent the dehydration illnesses.

The investigators will conduct a randomized controlled trial to examine the effectiveness of continuous home monitoring of fluid levels in a cohort of vulnerable older adult patients seen in the emergency care setting.

The goal of this randomized control trial is to examine the effectiveness of continuous home monitoring of fluid levels in older patients presenting to the emergency department for dehydration. The main questions it aims to answer:

1. Can a wearable device accurately determine the severity of dehydration at home and
2. can a wearable device and continuous feedback from the device change behavior in the outpatient setting that can lead to improved outcomes in the treatment of dehydration in the elderly?

Investigators will compare device readings, hydration diaries, vital signs, blood samples, return visits to the emergency department, and to see if feedback from the device decreases signs and symptoms of dehydration and changes home management of dehydration.

Participants will be asked to:

* wear the device and monitor hydration status
* record the amount of home hydration
* return in 7-10 days for reassessment of dehydration

The successful outcome of this study will include evidence for the effectiveness of the home, wearable hydration monitoring device, data necessary for the FDA 510(k) and related regulatory processes and substantial enhancements to both our knowledge of older adult needs and device functionality.

DETAILED DESCRIPTION:
Dehydration is common and costly: Dehydration is characterized by a decline in total body water. Dehydration is considered to be hypotonic when accompanying salt loss occurs and hypertonic if caused solely by water loss. Hypertonic dehydration is associated with mortality and severe short- term and long-term neurological sequelae. Annual costs of hospitalization primarily due to dehydration have been estimated at $1.36 billion. Approximately 17% of older adults hospitalized for dehydration die within 30 days, as often multiple organ systems are detrimentally affected by dehydration. Dehydration is not only widespread among older adults, but also an independent predictor of mortality. A number of studies have reported mortality rates associated with hypernatremia (a high sodium level that often accompanies dehydration) at greater than 40% and are commonly related to the underlying disease processes.

The cost of dehydration is twofold - one is the direct cost of dehydration on the patient and US healthcare; and second is its indirect effects as a comorbidity of another disease. For example, delirium is commonly caused by dehydration among older adults. In individuals with underlying dementia mild dehydration causes further cognitive impairment and possibly hallucinations, delusions, anxiety, and agitated behavior. Dehydration can also trigger other medical complications, such as infections, constipation, kidney stone formation, worsening aortic stenosis, valvular disease, adverse drug reactions, urinary tract infection, pneumonia, pressure ulcers, metabolic imbalance, uncontrolled diabetes, gastroenteritis, and some forms of cancer. According to an AHRQ study of the Nationwide Inpatient Sample (NIS) representing all patients in acute care hospitals, dehydration was diagnosed more commonly as a comorbidity than as a principal diagnosis. Dehydration was the second most common comorbidity, occurring in 14% of all hospitalizations. Thus, dehydration may contribute to the increase of medical costs in an indirect way. It may be a marker of the severity of the underlying disease, or it may add its own complications to those of the underlying disorder. Using direct costs alone, the potential annual U.S. savings from avoidable hospitalizations in these patients could have been as much as $1.14 billion. Dehydration is difficult to detect in real-time with traditional technologies: Primary reasons for the high prevalence of chronic dehydration among older adults are: (1) Older persons have metabolic and olfactory changes (2) medication regimens and disease consequences that can alter to their own fluid intake or the body's ability to maintain fluid levels (3) In older patients, access and maintenance of proper hydration is more difficult; for example, behavioral changes can include not wanting to drink to avoid incontinence in public and (4) traditional technologies do not present a simple, straightforward approach to measuring dehydration. Traditional measurement techniques are either obsolete, time consuming, inaccurate or not feasible. In our market survey, the investigators found that in current care settings care personnel check dehydration primarily through the use of visual signals or inferentially via blood-based indicators (e.g. sodium levels, creatinine). Skin elasticity checks, by pinching on hand or on the forehead, or checking the tongue (dry mouth), are still common. Not only are these methods are obsolete and inaccurate, care personnel are often skeptical of the results. Far too often, care personnel do not detect a dehydration in an older person until they are seriously ill and in need of emergency medical care.

Current Laboratory methods to detect dehydration: There are a few existing methods that can detect dehydration i.e. measure Total Body Water (TBW), intracellular water (ICW), and extracellular water (ECW). The tests involving urine, blood, or isotopic dilution are generally invasive, impractical or have not been adopted in either acute care or home settings. Furthermore, these tests can be difficult or impossible to repeat at regular intervals, precluding the opportunity to be used proactively and prevent dehydration. Total body composition machines on the market, which are based on bioimpedance measurement techniques have shown to be accurate and to deliver acceptable results in real time. However, a critical limitation of these devices is their size and thus ease of use in everyday setting. Other important barriers to using these devices for routine detection of dehydration include the electrode placement requirement (wrist to ankle or both hands and feet), equipment cost (>$10,000 per device) and no way of measuring the changes in the body fluids over time. To date, these devices are used almost exclusively in research or subspecialty care settings. Thus, even though these methods show promise of detecting dehydration in general, a simpler efficacious solution for measuring dehydration among community living older adults is highly desirable.

The D.R.INK device can detect falling hydration levels and alert individuals and care personnel to respond appropriately. Our proposed project will provide evidence for how our solution is transformative for inpatient, institutional care and community care settings alike by 1) making it user friendly to the population 2) ensuring its accuracy based on previously identified clinical and laboratory parameters 3) testing accuracy and effectiveness in a randomized observational setting and 4) determining how DRINK changes behavior and improve clinical outcomes. Thus the investigators expect that our real-time and accurate hydration monitoring device, has the potential to greatly reduce costly acute care among older adults. The band is expected to not only improve the overall quality of life older adults but also reduce the morbidity and mortality, by enabling the proactive detection of an avoidable condition: dehydration.

A key advantage of the DRINK technology over other methods is that the device can detect changes in fluid levels by collecting longitudinal data within person at regular intervals outside of the clinical settings. In addition to the immediate benefits in our proposed work the investigators expect a wide range of future applications and the ability to uncover tremendous health insights.

This project aims to:

1. Examine the effectiveness of continuous home monitoring of fluid levels. Hypothesis 1: A wearable hydration device improves recovery after acute care for dehydration Hypothesis 2: A wearable hydration device reduces acute negative health events among a vulnerable population of older adults at risk for dehydration.
2. Combine clinical expertise and results from outcomes measurement to define measurement indicators, propose clinically actionable thresholds, safety guidelines and improved visualizations for patients and care teams.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged 55 and over
* rresenting to the emergency department
* clinical suspicion of dehydration
* treatment of dehydration/syncope with fluid resuscitation
* English speaking

Exclusion Criteria:

* Refusal or inability to give informed consent,
* severe clinical symptom requiring escalation of care beyond fluid resuscitation (ex. vasopressors, invasive blood pressure monitoring)
* presumed/confirmed diagnosis of syncope secondary to a non-dehydration cause (ex. arrhythmia, stroke, pulmonary embolism, sepsis, valvular heart disease)
* inability to lay flat for the test
* body weight greater than 350 lbs
* inability to fit measurement devices around the participant wrist
* abnormal bodily fluid retention (lymphedema, ascites, pleural effusions, peripheral edema)
* neuromotor disorders
* current congestive heart failure exacerbation or heart attack/myocardial infarction
* any implantable electronic devices
* skin on limbs in poor condition (excessively, dry or rough or abrasions or wounds that would preclude application of electrode adhesive)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Average daily fluid intake in mL | 10 days
  The average daily fluid intake over 10 days as determined by a standardized Drink Diary

SECONDARY OUTCOMES:
Level of total body water after 10 days | 10 days
  Total body water after 10 days will be determined by the wearable dehydration device
Midpoint Clinical symptoms of dehydration | 5 days
  Midpoint telehealth visit reports of syncope, dizziness, feeling of confusion, increased thirst, reported decreased urinary output, feeling fatigued
End of Study Report of Dehydration | 10 days
  Any reported syncope, dizziness, feeling of confusion, increased thirst, reported decreased urinary output, feeling fatigued.
End of Study Visit Heart Rate (beats per minute) | 10 days
  HR >100 would be considered abnormal
End of Study Visit Blood Pressure | 10 days
  Systolic and diastolic blood pressure (mmHg)
End of Study Visit Orthostatic Vital Signs | 10 days
  HR and BP upon standing and sitting. HR rate of change greater than 30 bpm or symptoms of dizziness would be considered positive
End of Study Visit Serum Osmolality | 10 days
  measured in mOsm/kg
End of Study Visit Serum Sodium | 10 days
  measured in mEq/L
End of Study Visit Serum Creatinine | 10 days
  measured in mg/dL
End of Study Visit Glomerular Filtration Rate | 10 days
  estimated GFR in milliliters per minute per body surface area

CONTACTS AND LOCATIONS:
Overall Officials: Jospeh S Piktel, MD, Principal Investigator — MetroHealth System, Ohio

IPD SHARING:
Plan to Share IPD: No
Summary data will be available but we may not share individual data due to concern for patient privacy